CLINICAL TRIAL: NCT05991609
Title: Establishing the Metabolic and Nutritional Requirements of Individuals With Extreme Body Morphology
Brief Title: Extreme Morphology and Metabolic Health
Status: Active, not recruiting | Type: Observational
Sponsor: University of Bath (Other)
Collaborators: University of Bristol (Other)
Responsible Party: Principal Investigator, James Betts, Professor, University of Bath
Other Study IDs: 321662
Record Dates: First submitted 2023-07-20; First posted 2023-08-14 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Skeletal Dysplasia
Keywords: Morphology; Skeletal dysplasia; Metabolism
MeSH Terms: conditions — Mucopolysaccharidosis IV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Buffy coat layer from blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Individuals with extreme body size: Any individual with a form of skeletal dysplasia, or extremely small or large body size.

SUMMARY:
Researchers at the University of Bath are investigating the metabolism of individuals with extreme body size, including those with skeletal dysplasia (commonly known as dwarfism), to manage health risks such as heart disease. By better understanding how body size could change how the body processes food, or how being bigger or smaller may influence eating habits, healthy living guidelines to tackle issues such as obesity and overweight in these populations can be improved. With help from expertise in the psychology field, this research will also investigate whether the mental health of these individuals has been affected by their size. On the whole, this study will involve one 24-hour visit to a research laboratory at the University of Bath, followed by a 2-week monitoring period to capture 'normal' physical activity and eating routines.

DETAILED DESCRIPTION:
After signing informed consent to take part in the study, participants will be asked to complete a health entry criteria questionnaire, including a physical activity readiness questionnaire and Eating Disorder Examination Questionnaire, to confirm eligibility. Participants will also be required to complete a health questionnaire for administration of anaesthetic as part of the biopsy procedure. Individuals who are very small or very big (without skeletal dysplasia) will be asked to attend the laboratory for a pre-trial screening as an additional eligibility criterion. This will involve measuring height, body mass, and standing on a specialised scale (bioelectrical impedance scale) which estimates how much muscle and fat someone has. If it is suspected that the participant meets the stated fat-free mass criteria, a complete a full body Dual Energy X-ray Absorptiometry (DEXA) scan to assess body composition more accurately will be completed. This involves lying flat on a bed for ~7 minutes and resting whilst the scan takes place. The research team will then inform the participant after analysing the scan results if they are eligible and can continue with the study.

All participants deemed eligible who are able and willing to take part will be invited to attend the University of Bath Human Physiology Laboratory for the full trial.

On day 1, prior to attending the University of Bath participants will be asked to eat a standardised diet of a cereal breakfast, and a supermarket purchased sandwich, drink and snack meal deal for lunch, with self-selected quantities. Participants will ideally be fasted for 4-5 hours before arrival (~17:00).

Upon arrive at the University, individuals with skeletal dysplasia will also be asked to complete the health entry criteria questionnaire and physical activity readiness questionnaire to ensure eligibility. It is important that participants let the researchers know of any medical conditions or any change in circumstance since signing up. All information is strictly confidential.

The research team will first take measurements of height, body mass, waist and hip circumference, abdomen diameter (distance from your front to back), sitting height and blood pressure. Early into the visit, participants will also be briefed on collecting urine into provided containers. Individuals with skeletal dysplasia will then have a Dual Energy X-ray Absorptiometry (DEXA) scan to assess body composition. All participants will also have a Peripheral Quantitative Computed Tomography (pQCT) scan which involves placing one leg into a round scanner to assess the tissues in your leg e.g., bone, muscle and fat (as if the image were a slice). The scan requires you to keep your leg still for ~10 minutes.

Participants will then be asked to rest in a bed and relax. In a seated position, participants will complete a lung function test at rest which requires blowing into a specialised device through a mouthpiece. Following this, after lying down and being briefed on the procedure, a trained member of staff will take a fat tissue biopsy from the abdomen to analyse genes and proteins in the cells. The fat biopsy involves inserting a needle with suction just below the skin to extract the cells and will be performed under local anaesthetic. This procedure may cause a bruise for up to 7 days. Following on from this, a muscle biopsy will be taken from the quadriceps (large muscle on the front of the thigh) to again measure genes and proteins as well as signalling pathways involved in our metabolism. The needle is inserted just inside the muscle and 2/3 snips of tissue are collected. The research team will provide information and equipment for aftercare of the biopsy sites to prevent infection after participants leave the laboratory.

Participants will then be provided with a hot meal for dinner. This will be a standard portion of Sainsbury's Love Your Veg! Lentil Cottage Pie (400 g, serves 1). Prior to turning the lights out at 22:00, participants will be fitted with sleep monitoring kit known as polysomnography. The equipment includes an abdominal and chest pressure sensing band, a nasal cannula and some sticky sensors placed directly on the skin.

On the morning of day 2, a researcher will wake the participant at 07:00. Using a mouthpiece (alike to a snorkel) and nose clip, expired air at rest will be collected for 20 minutes to calculate how much energy is burnt at rest. Participants will also be asked to give a breath sample into a small glass tube through a straw (this is related to a tracer method explained below). Body mass will be measured again after the participant has an opportunity to use the bathroom.

Once settled back in bed, a trained member of staff will insert a cannula (small plastic tube) into a vein on the back of the participant's hand or forearm. This will stay in place for the remainder of the day and allows repeated blood samples to be taken throughout the following tests. For participants with skeletal dysplasia, the genetic material found in cells will be taken out of the first blood sample and later analysed to confirm a correct diagnosis of achondroplasia. Participants will be asked to place the hand in a warm box set at 55°C which helps blood flow and makes taking samples easier for the research team. All participants will then be asked to complete a series of appetite questions, a portion selection task, and blood pressure will be taken.

When the hand is warm and initial appetite tasks are completed, participants will be provided with a sugary drink and asked to finish it within 5 minutes. The drink will also contain a sugar tracer which is stable and safe-to-consume. This allows the research team to assess how the drink is being processed by the body in real time. For a few individuals from each 'subgroup' (achondroplasia, skeletal dysplasia, extremely large body size, and extremely small body size), a different tracer called acetate will be added to the drink which will help with some calculations of how the body processes the sugar. Blood samples (10 mL) will be drawn from the cannula every 15 minutes for the first hour, and 30 minutes for the next two hours. At these same intervals, the participant will be asked to blow into a small tube using a straw to assess the appearance of the tracer on the breath (an indicator of how much sugar is being burnt from the drink, as opposed to the body's sugar stores, hence the need for a baseline sample). Participants will also be asked to complete the appetite questions and portion selection task whenever a blood sample is drawn. At 60, 120 and 180 minutes, a one 5-minute sample of air will be collected just as upon waking, and blood pressure will be measured on the hour. In between samples the participant may also complete a series of questionnaires regarding mental health (optional).

At 11:00, participants will be presented with another appetite task and then a lunch meal (pesto pasta with cheese, and a glass of orange juice) to consume within 20-minutes. A few additional appetite questions will be asked pre- and post- meal consumption. The following 3 hours will be similar to before, with regular appetite scales to complete, and blood samples drawn every 15 minutes for the first hour, and 30 minutes for the next two hours. At 60, 120 and 180 minutes, one 5-minute breath sample and a smaller tracer breath sample through the straw will be collected, and blood pressure recorded.

Participants will then be asked to complete a short treadmill test to calibrate the activity monitor by wearing a heart rate monitor on a chest strap whilst walking. Five 3-minute incremental stages will be calculated based on the participants 'normal' self-selected walking speed. During the final minute of each stage, a one-minute breath sample will be collected and heart rate recorded. A breath sample into a tracer collection tube will also be obtained at the end of each exercise stage. Whilst on the treadmill, participants will be asked to describe how difficult the exercise stages feel. If the fastest speed has not exceeded 'hard' exercise, the researcher will ask if the participant feels able to complete a final stage at a higher intensity (not exceeding a rating of perceived exertion of 15) to assist calibration of the activity monitor. Within 30 seconds of finishing on the treadmill one final blood sample will be drawn from the cannula before removing it.

On leaving the lab, participants will be provided with an activity monitor, a motion watch, a food diary (either on a mobile app or paper copy), and food and body weight scales. A small device to continuously measure blood sugar levels will also be fitted to the back of the arm. The device is inserted with a very small needle which is then removed, leaving only the patch with a small probe in the arm. The research team will instruct participants on how to wear the activity monitor on the chest and ask that participant wear this at all times other than when swimming or bathing, and record food intake for 14-days. During this time, participants will be asked to weigh themselves first thing in the morning and last thing at night, as well as recording sleep times and quality.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 years or over
* Any diagnosed form of skeletal dysplasia (i.e., extreme proportionate or disproportionate short stature)
* Individuals without skeletal dysplasia but presenting with extreme body morphology, defined as: individuals with extreme large body morphology (males >75 kg fat-free mass and females >57.25 kg fat-free mass), or males and females with extreme small body morphology (<47.4 kg fat-free mass).

Exclusion Criteria:

* Any reported condition, behaviour or reported use of substances which may pose undue personal risk to the participant or introduce bias into the study, except for any which are ubiquitous in society and so would be equally distributed between groups and/or therefore relevant to generalisation (e.g., statins, caffeine, GLP-1 agonists).
* Females who are pregnant or lactating
* Individuals with a diagnosed history of eating disorders (e.g., anorexia)
* Individuals with known bleeding disorders (exclusion for biopsies only)
* Individuals with known allergy or intolerance to lidocaine
* Inability to read or speak English, or otherwise to consent to procedures
* Individuals who are not weight stable (i.e., >3 kg change in body mass in past 3 months)

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with extreme body size or proportions.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2023-06-17 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2035-09-28 (Estimated)

PRIMARY OUTCOMES:
Glucose incremental area under the curve during the oral glucose tolerance test | 3 hours
  Difference in blood glucose incremental area under the curve between individuals with skeletal dysplasia, and extremely small and large body size.

SECONDARY OUTCOMES:
Fasted blood glucose concentration | Baseline
Fasted blood insulin concentration | Baseline
Insulin response to oral glucose tolerance test | 3 hours
  Incremental area under the curve of blood insulin after oral glucose tolerance test
C-Peptide response to oral glucose tolerance test | 3 hours
  Incremental area under the curve of blood C-Peptide after oral glucose tolerance test
Regulatory hormone response to oral glucose tolerance test | 3 hours
  Incremental area under the curve of regulatory hormones e.g. ghrelin after oral glucose tolerance test
Glycaemic response to mixed meal tolerance test | 3 hours
  Incremental area under the curve of blood glucose after mixed meal tolerance test
Insulin response to mixed meal tolerance test | 3 hours
  Incremental area under the curve of blood insulin after mixed meal tolerance test
C-Peptide response to mixed meal tolerance test | 3 hours
  Incremental area under the curve of blood C-Peptide after mixed meal tolerance test
Regulatory hormone response to mixed meal tolerance test | 3 hours
  Incremental area under the curve of regulatory hormones e.g. ghrelin after mixed meal tolerance test
Resting metabolic rate | Baseline
Substrate oxidation during oral glucose tolerance test | 3 hours
  Total fat and carbohydrate oxidation
Substrate oxidation during mixed meal tolerance test | 3 hours
  Total fat and carbohydrate oxidation
Exogenous carbohydrate oxidation | 7 hours
  Time course for whole-body exogenous carbohydrate using stable isotope methodology
Fasting muscle glycogen concentration | Baseline
  Difference between individuals with skeletal dysplasia, extremely small and large body morphology.
Non-oxidative glucose disposal | 7 hours
  Difference in exogenous carbohydrate consumption and exogenous carbohydrate oxidation
Continuous interstitial glucose concentration | 10 days
Adipose tissue markers of insulin signalling | Baseline
Adipose tissue markers of glucose metabolism | Baseline
Skeletal muscle markers of insulin signalling | Baseline
Skeletal muscle markers of glucose metabolism | Baseline
Fasted concentration of systemic adipokines (e.g., adiponectin, resistin, leptin etc.) | Baseline

OTHER OUTCOMES:
Height | Baseline
  Metres
Body mass | Baseline
  Kilograms
Change in body mass over 14 days of free-living monitoring | 14 days
  Kilograms
Waist:Hip ratio | Baseline
Sagittal abdominal diameter | Baseline
  Centimeters
Blood pressure | 6 hours
  mmHg
Intracellular markers and signalling pathways related to carbohydrate metabolism in adipose tissue | Baseline
  Comparing adipose tissue between skeletal dysplasia, extremely small and large groups
Intracellular markers and signalling pathways related to carbohydrate metabolism in skeletal muscle | Baseline
  Comparing muscle tissue between skeletal dysplasia, extremely small and large groups
Full blood lipid profile | 7 hours
  Blood analysed and compared between skeletal dysplasia, extremely small and large groups
Fasted markers of chronic low-grade inflammation | Baseline
  Blood analysed and compared between skeletal dysplasia, extremely small and large groups
FGFR protein expression and signalling pathway exploration | Baseline
  Muscle tissue analysed and compared between skeletal dysplasia, extremely small and large groups
24-hour protein oxidation | 24 hours
  Grams per minute
Genotype- FGFR3 mutation (skeletal dysplasia group only) | Baseline
  Assessed from buffy coat layer
Panel of female sex hormones | Baseline
  To verify menstrual cycle phase
DEXA bone mineral density | Baseline
DEXA fat mass | Baseline
DEXA fat-free mass | Baseline
pQCT - muscle cross-sectional area | Baseline
pQCT - tissue density | Baseline
pQCT - bone geometry | Baseline
Assessment of eating behaviour | Baseline
  The Three Factor Eating Questionnaire
Visual analogue scale appetite ratings | 6 hours
Portion selection task | 6 hours
Polysomnography profile | Baseline
Daily self-reported energy intake during free-living monitoring | 14 days
  Daily self-reported energy intake using Nutritics Libro Application
Daily free-living physical activity energy expenditure | 14 days
  Daily free-living physical activity measured by Actiheart monitor
Free-living sleep quality | 14 days
Free-living sleep duration | 14 days
Free-living light exposure | 14 days
Diet induced thermogenesis | 14 days
  Calculated from self-reported energy intake
Heart rate during exercise | 15 minutes
  Beats per minute
Rate of perceived exertion during exercise | 15 minutes
  BORG scale
Energy expenditure during exercise | 15 mins
  Substrate oxidation during walking exercise
Mental health assessment | Baseline
  Validated questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: James A Betts, PhD, Principal Investigator — University of Bath
Locations (1):
- University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: No